CLINICAL TRIAL: NCT06739343
Title: Comparison of Phaco-Trabeculectomy Versus Combined Manual Small Incision Cataract Surgery with Trabeculectomy in Patients with Coexisting Cataract and Glaucoma At ECWA Eye Hospital, Kano, Nigeria
Brief Title: Comparison of Phaco-Trabeculectomy and MSICS-Trab in Cataract and Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emeka John Dingwoke (Other)
Collaborators: Ahmadu Bello University Teaching Hospital (Other)
Responsible Party: Sponsor-Investigator, Emeka John Dingwoke, Director, UNESCO International Centre for Biotechnology, Nigeria
Organization: UNESCO International Centre for Biotechnology, Nigeria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECWA/HREC/004/2022
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cataract; Glaucoma
Keywords: Cataract; Glaucoma; Phaco-Trabeculectomy; MSICS-Trabeculectomy; Intraocular Pressure; Visual Acuity; ECWA Eye Hospital; Surgical Outcomes; Combined Surgery; Ophthalmology
MeSH Terms: conditions — Cataract; Glaucoma

STUDY DESIGN:
Intervention Model Description: This study follows a parallel group design, where eligible participants are randomly assigned to one of two independent intervention arms: the Phaco-Trabeculectomy group or the MSICS-Trabeculectomy group. Each group receives a distinct surgical intervention, and participants remain in their assigned groups throughout the study duration. Outcomes are measured and compared between the two groups to evaluate the relative effectiveness and safety of the interventions.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PHACO-Trabeculectomy Group (Active Comparator): Participants in this group underwent Phaco-Trabeculectomy, a combined surgical procedure that involves phacoemulsification (modern cataract extraction technique) and trabeculectomy (a glaucoma filtration surgery). This procedure is designed to address both cataract removal and intraocular pressure (IOP) reduction in a single surgery.
  Interventions:
  Phacoemulsification: Ultrasound-based cataract removal. Trabeculectomy: Creation of a filtration bleb to lower IOP.
  Interventions: Procedure: PHACO-Trabeculectomy; Procedure: MSICS-Trabeculectomy
- MSICS-Trabeculectomy Group (Active Comparator): Participants in this group underwent Manual Small Incision Cataract Surgery (MSICS) combined with trabeculectomy. This procedure, which uses a manual technique for cataract extraction, is often more cost-effective and suitable for resource-limited settings while also addressing IOP reduction.
  Interventions:
  Manual Small Incision Cataract Surgery (MSICS): A manual extracapsular cataract extraction technique.
  Trabeculectomy: Same filtration procedure as in the Phaco-Trabeculectomy group to manage glaucoma.
  Interventions: Procedure: PHACO-Trabeculectomy; Procedure: MSICS-Trabeculectomy

INTERVENTIONS:
Procedure: PHACO-Trabeculectomy — Phaco-Trabeculectomy is a combined surgical procedure that integrates phacoemulsification, a modern cataract extraction technique using ultrasound, with trabeculectomy, a glaucoma filtration surgery. This intervention is distinguished by its precision, minimal incision size, and suitability for patients with coexisting cataract and glaucoma. Phacoemulsification efficiently emulsifies and aspirates the cataract through a small incision, while trabeculectomy creates a filtration bleb to lower intraocular pressure (IOP). This combination allows for simultaneous management of both conditions, particularly in cases where phacoemulsification is preferred for cataract extraction.
Procedure: MSICS-Trabeculectomy — Manual Small Incision Cataract Surgery (MSICS) with Trabeculectomy is a cost-effective, combined surgical approach involving a manual technique for cataract removal alongside glaucoma filtration surgery. MSICS utilizes a larger incision than phacoemulsification, allowing for the manual extraction of the cataract nucleus. This procedure is particularly advantageous in resource-limited settings where phacoemulsification equipment may not be available. The trabeculectomy component is the same as in the PHACO-Trabeculectomy intervention, providing effective IOP reduction through the creation of a filtration bleb.

SUMMARY:
The goal of this interventional study is to compare the outcomes of two surgical techniques, Phaco-Trabeculectomy and Manual Small Incision Cataract Surgery (MSICS) with Trabeculectomy, in patients with coexisting cataract and glaucoma at ECWA Eye Hospital, Kano, Nigeria. The study aims to evaluate which technique offers better intraocular pressure (IOP) control, visual acuity improvement, and complication rates postoperatively.

The main questions the study seeks to answer are:

Does Phaco-Trabeculectomy provide superior IOP control compared to MSICS-Trabeculectomy in patients with coexisting cataract and glaucoma? Which technique is associated with fewer postoperative complications? How do the visual outcomes compare between the two techniques? Participants will be randomly assigned to undergo one of the two surgical techniques based on a predefined protocol. Data will be collected on intraoperative and postoperative parameters, including IOP, visual acuity, and the incidence of complications, with follow-ups extending over a 12-month period.

This study aims to provide evidence to guide clinicians in selecting the most effective and safe surgical approach for managing patients with cataract and glaucoma in resource-limited settings.

DETAILED DESCRIPTION:
Background and Rationale Cataract and glaucoma are two of the leading causes of preventable blindness globally, presenting significant public health challenges, particularly in resource-limited settings such as Nigeria. The coexistence of cataract and glaucoma complicates surgical management, as cataract surgery alone may improve visual acuity but is insufficient to achieve long-term control of intraocular pressure (IOP) in glaucoma patients.

Combined surgical procedures, such as Phaco-Trabeculectomy and Manual Small Incision Cataract Surgery (MSICS) with Trabeculectomy, have been adopted to address these dual ocular conditions in a single intervention. However, evidence comparing the efficacy, safety, and long-term outcomes of these two approaches remains limited, particularly in Sub-Saharan Africa. This study seeks to bridge this critical gap in clinical evidence by generating region-specific data to optimize surgical decision-making for patients with coexisting cataract and glaucoma.

ECWA Eye Hospital, Kano, a tertiary eye care center in Nigeria renowned for its excellence in ophthalmology, provides the ideal setting for conducting this interventional study.

Study Objectives

This study aims to:

Determine whether Phaco-Trabeculectomy or MSICS-Trabeculectomy offers superior intraocular pressure (IOP) control in patients with coexisting cataract and glaucoma.

Compare the visual acuity outcomes between the two surgical techniques. Evaluate and compare the incidence of postoperative complications, such as bleb failure, hypotony, and infection.

Assess patient satisfaction and quality of life using validated questionnaires.

Study Design

This is a randomized, parallel-group, interventional study conducted over a 12-month follow-up period. Eligible participants are randomized into two arms using a block randomization approach to ensure balanced allocation:

Phaco-Trabeculectomy Group MSICS-Trabeculectomy Group Randomization minimizes selection bias and ensures comparability of baseline characteristics between groups.

Key Surgical Interventions Phaco-Trabeculectomy This procedure integrates phacoemulsification, a modern cataract extraction technique, with trabeculectomy to achieve IOP control.

A 3.2 mm corneal incision is made for ultrasonic emulsification and aspiration of the cataract.

A trabeculectomy is performed to create a filtration bleb, facilitating aqueous humor drainage.

This method is precise, minimally invasive, and well-suited for modern ophthalmic practice.

MSICS-Trabeculectomy This procedure combines manual extracapsular cataract extraction with trabeculectomy and is particularly advantageous in resource-limited settings.

A fornix-based conjunctival flap is raised, and a larger manual incision is made to remove the cataract nucleus.

Trabeculectomy is performed using the same technique as in the Phaco-Trabeculectomy group.

The MSICS-Trabeculectomy approach is practical, cost-effective, and suitable for environments where phacoemulsification equipment is unavailable.

Postoperative Management

Standardized postoperative care includes:

Administration of topical corticosteroids, antibiotics, and anti-glaucoma medications to reduce inflammation, prevent infection, and manage IOP.

Follow-up visits conducted on day 1, week 1, months 1, 3, 6, and 12 to assess clinical outcomes and monitor for complications, including hypotony, bleb failure, and infection.

Bleb morphology is evaluated using validated grading systems, while patient satisfaction and quality of life are assessed using standardized questionnaires.

Data Collection and Analysis

Data on surgical outcomes, including IOP, visual acuity, and postoperative complications, are systematically collected at predefined intervals. Statistical tools are employed for comparative analysis:

Continuous variables such as IOP and visual acuity are analyzed using paired and unpaired t-tests.

Categorical variables, including complication rates, are analyzed using chi-square tests and logistic regression models.

Results will be presented as mean ± standard deviation for continuous variables and as percentages for categorical variables.

Significance of the Study

This study provides a direct comparative analysis of Phaco-Trabeculectomy and MSICS-Trabeculectomy in a Sub-Saharan African context. By evaluating clinical efficacy, cost-effectiveness, and patient-reported outcomes, the findings will:

Inform clinical practice by identifying the optimal surgical approach for managing coexisting cataract and glaucoma.

Address regional gaps in evidence-based ophthalmic care, particularly in resource-limited settings.

Serve as a foundation for further studies exploring long-term surgical outcomes and innovations in glaucoma-cataract management.

Novel Contributions

This study is one of the first to comprehensively evaluate two combined surgical techniques in a Sub-Saharan African population. Its strengths include:

Rigorous randomization to ensure unbiased comparisons. Systematic data collection at predefined intervals over 12 months. Use of validated tools for assessing bleb morphology, complications, and patient satisfaction.

By bridging the gap in clinical evidence, this study has the potential to improve surgical decision-making, enhance patient outcomes, and guide ophthalmic care strategies in resource-constrained settings.

Conclusion This interventional study will provide critical insights into the comparative effectiveness and safety of Phaco-Trabeculectomy and MSICS-Trabeculectomy for managing coexisting cataract and glaucoma. Its findings are expected to have significant implications for ophthalmic practice in Nigeria and other resource-limited regions, ultimately contributing to the prevention of avoidable blindness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years.
* Patients diagnosed with coexisting cataracts and primary open-angle glaucoma.
* Patients who have provided informed consent to participate in the study.

Exclusion Criteria:

* Patients with angle-closure glaucoma.
* Patients with secondary glaucoma or glaucoma-associated ocular or systemic anomalies.
* Patients with a history of ocular surgeries, such as trabeculectomy, cataract surgery, or other glaucoma surgeries.
* Patients with corneal or anterior segment diseases that could impede detailed examination (e.g., scleritis, bullous keratopathy, corneal scarring, corneal degenerations, or uveitis).
* Patients with posterior segment diseases affecting visual interpretation (e.g., diabetic retinopathy, hypertensive retinopathy, high axial myopia, retinal detachment, vitreous hemorrhage, macular degeneration, central retinal vein occlusion, or sickle cell retinopathy).
* Patients unwilling to provide voluntary informed consent or those who chose to withdraw from the study at any point.
* Patients with only one functional eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Intraocular Pressure (IOP) | Baseline, Day 1, Week 1, Month 1, Month 3, Month 6, and Month 12 post-surgery. To determine the relative effectiveness of the two surgical techniques in managing glaucoma-related elevated IOP.
  The primary outcome measure is the change in intraocular pressure (IOP) from baseline to 12 months postoperatively. IOP will be measured using the Goldmann Applanation Tonometer, the gold standard for IOP measurement. Measurements will be recorded in millimeters of mercury (mmHg).
  The change in intraocular pressure (IOP) will reflect the effectiveness of the surgical intervention in controlling IOP over time. Lower IOP values within the normal range (10-21 mmHg) indicate successful pressure regulation and better surgical outcomes, reducing the risk of glaucoma progression. Conversely, persistently elevated IOP values may suggest surgical failure
  The changes in IOP will be compared between the Phaco-Trabeculectomy and MSICS-Trabeculectomy groups to assess the efficacy of each surgical technique in controlling intraocular pressure over the study duration.

SECONDARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) | Baseline, Month 1, Month 3, Month 6, and Month 12 post-surgery
  Secondary outcomes include the improvement in best-corrected visual acuity (BCVA), measured using the Snellen chart.
  BCVA is expressed in logMAR units, with lower logMAR values reflecting better visual acuity.
  For instance, a logMAR of 0.1 corresponds to good vision (6/7.5), while higher values indicate worsening acuity.
Postoperative Complications | Day 1, Week 1, Month 1, Month 3, Month 6, and Month 12 post-surgery.
  Hypotony will be recorded and compared between the two groups. Hypotony: Defined as intraocular pressure (IOP) <5 mmHg, will be measured using the Goldmann tonometer (unit: mmHg). Lower IOP values below 5 mmHg indicate hypotony. Higher IOP values within the normal range (10-21 mmHg) reflect better intraocular pressure control and stable ocular function.
Bleb Function | Month 1, Month 3, Month 6, and Month 12 post-surgery
  Assessment of the filtration bleb's functionality will be done using the Indiana Bleb Appearance Grading Scale (IBAGS). This standardized grading system evaluates bleb vascularity (graded V0-V4).
  Lower grades (V0-V1) indicate minimal or no vascularity, suggesting a healthy and functional bleb, which is favorable for successful aqueous humor drainage and intraocular pressure control. Higher grades (V3-V4) reflect increased vascularity, which may signal inflammation.

OTHER OUTCOMES:
Patient-Reported Satisfaction | Month 3 and Month 12 post-surgery
  Patient satisfaction and quality of life postoperatively will be assessed using Visual Function Questionnaire (VFQ-25).
  Standardization:
  VFQ-25: Measures visual function and its impact on daily activities. Scores range from 0 to 100, with higher scores indicating better visual function and quality of life.
Patient-Reported Quality of Life | Day 1, Week 1, Month 1, Month 3, Month 6, and Month 12 post-surgery.
  Quality of life in glaucoma patients as assessed using the Glaucoma Quality of Life-15 (GQL-15). Scores range from 0 to 75, where lower scores reflect fewer difficulties and better quality of life.
Duration of Surgery | Intraoperative (30-90 minutes). The intraoperative period spans the duration of the surgical intervention, beginning with anesthesia administration and ending upon completion of the procedure.
  The time taken to complete each surgical procedure (Phaco-Trabeculectomy vs. MSICS-Trabeculectomy) will be recorded to assess operational efficiency.
Cost Analysis | Throughout the study duration (baseline, 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months). Data will be collected at these specific time points to evaluate outcomes across the study period.
  The overall cost of each procedure will be analyzed to evaluate cost-effectiveness.
  Costs will be recorded per patient and reported as the mean cost per procedure for the Phaco-Trabeculectomy and MSICS-Trabeculectomy groups.
  Units of Measure: Costs will be expressed in Nigerian Naira (NGN), and comparative analysis will highlight the cost differences and cost-effectiveness between the two surgical techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Mayor Orezime Atima, FWACS, Study Chair — ECWA Eye Hospital, Kano
Locations (1):
- ECWA Eye hospital, Kano, Kano State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) related to primary and secondary outcome measures will be shared with researchers upon reasonable request. Data will be anonymized and made available through a secure repository following approval of a data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date: 6 months after the publication of study results End Date: Available for 5 years following publication.
Access Criteria: Who Will Have Access:
  Qualified researchers affiliated with academic institutions, research organizations, or healthcare entities will be eligible to request access.
  What Will Be Accessible:
  De-identified individual participant data (IPD) relevant to primary and secondary outcome measures, along with supporting documentation such as the study protocol, statistical analysis plan, and informed consent templates.
  How Access Will Be Granted:
  Interested researchers must submit a formal request including a detailed research proposal outlining the intended use of the data. Requests will be reviewed by a data-sharing committee or principal investigator. Approved researchers will be required to sign a data-sharing agreement ensuring data confidentiality, compliance with ethical guidelines, and appropriate use of the data.
  Access Mechanism:
  Data will be shared via a secure online repository or data-sharing platform. Approved researchers will receive time-limited credentials to access the data

REFERENCES:
- [Derived] Munaje MI, Aribaba OT, Atima MO, Idakwo U, Pam JD, Dingwoke EJ, Gandi NB. Phaco-trabeculectomy versus MSICS-trabeculectomy for coexisting cataract and glaucoma: visual and IOP outcomes from a randomized trial in Nigeria. BMC Ophthalmol. 2025 Nov 5;25(1):621. doi: 10.1186/s12886-025-04482-1. PMID 41194003